CLINICAL TRIAL: NCT01026181
Title: Phase II Study of Comparing Outcomes of Laparoscopic Sleeve Gastrectomy, Laparoscopic Roux-en-Y Gastric Bypass and Laparoscopic Gastric Banding to Treat Morbid Obesity
Brief Title: Gastric Procedures for Obesity
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Principal Investigator, Shahzeer Karmali, BSc, MD, FRCSC, University of Alberta
Other Study IDs: Pro00002425
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Results first posted 2017-10-03 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-05

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- LSG: Laparoscopic Sleeve Gastrectomy
- LRYGB: Laparoscopic Roux-en-Y Gastric Bypass
- LAGB: Laparoscopic Adjustable Gastric Banding

SUMMARY:
This is a prospective case series study; all morbidly obese patients that need surgical management in Royal Alexandra Hospital will be provided 3 surgical options: Laparoscopic Sleeve Gastrectomy (LSG), laparoscopic Roux-en-Y gastric bypass (LR-en-Y), and laparoscopic gastric banding (LGB), safety and effectiveness will be compared among the 3 groups. The outcome measures will be percentage of excess weight loss, BMI, operative time, hospital stays, complications and improvement of comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* morbid obese patients aged from 18-65,
* BMI > 40 kg/m2 or BMI> 35 kg/m2 with severe comorbidities: diabetes, sleep apnea, hypertension etc.

Exclusion Criteria:

* psychiatric illness,
* substance abuse,
* previous gastrointestinal surgery, and
* any patient who transfers from laparoscopic to convention procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Morbidly obese patients aged from 18 to 65.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2008-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Laparoscopic Sleeve Gastrectomy: Patient who had Laparoscopic Sleeve Gastrectomy for their morbid obesity
- Laparoscopic Roux-en-Y Gastric Bypass: Patients who had Laparoscopic Roux-en-Y Gastric Bypass for their morbid obesity
- Laparoscopic Adjustable Gastric Banding: Patients who had Laparoscopic Adjustable Gastric Banding for their morbid obesity
Period: Overall Study
Arm/Group | Laparoscopic Sleeve Gastrectomy | Laparoscopic Roux-en-Y Gastric Bypass | Laparoscopic Adjustable Gastric Banding
Started | 51 | 51 | 48
Completed | 51 | 51 | 48
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- LSG (Lap SG): Laparoscopic Sleeve Gastrectomy
- Total: Total of all reporting groups
Arm/Group | LSG (Lap SG) | LRYGB | LAGB | Total
Number analyzed (Participants) | 51 | 51 | 48 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (9.6) | 41.9 (8.4) | 43.1 (10.3) | 43.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 41 | 45 | 131
  Male | 6 | 10 | 3 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  race: white race | 46 | 51 | 44 | 141
  race: other race | 5 | 0 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Change of body weight in Kilograms measured at follow-up visits two year after surgery
Time Frame: baseline to 2-year postoperation
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Laparoscopic Sleeve Gastrectomy | Laparoscopic Roux-en-Y Gastric Bypass | Laparoscopic Adjustable Gastric Banding
Number analyzed (Participants) | 51 | 51 | 48
kg | -21.4 (16) | -36.6 (19.5) | -7.0 (9.7)

2. Primary Outcome: Change in BMI
Description: Patients' weight and height were measured at follow up visit 2 years post operation.
  BMI was calculated using the formula: weight (kg)/height(meter)^2
Time Frame: from baseline to 2-year postoperation
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Laparoscopic Sleeve Gastrectomy | Laparoscopic Roux-en-Y Gastric Bypass | Laparoscopic Adjustable Gastric Banding
Number analyzed (Participants) | 51 | 51 | 48
kg/m^2 | -7.6 (5.7) | -13.0 (6.6) | -2.6 (3.5)

ADVERSE EVENTS:
Time Frame: 2 year after surgery.
Description: Adverse events were classified according to a modified Clavien-Dindo surgical complications system, focusing on grade III or higher. All reported adverse events required intervention, admission, or re-operation. Other non-serious adverse events were not collected/assessed.
Arm/Group | Laparoscopic Sleeve Gastrectomy | Laparoscopic Roux-en-Y Gastric Bypass | Laparoscopic Adjustable Gastric Banding
Serious Adverse Events (participants affected / at risk) | 5/51 | 10/51 | 7/48
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laparoscopic Sleeve Gastrectomy (N=51) | Laparoscopic Roux-en-Y Gastric Bypass (N=51) | Laparoscopic Adjustable Gastric Banding (N=48)
gastrointestinal/staple line leak (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0)
gastrointestinal/staple line bleed (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
anastamotic ulcer (Surgical and medical procedures) | 0 (0) | 3 (3) | 0 (0)
stricture (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
band slippage (Surgical and medical procedures) | 0 (0) | 0 (0) | 6 (6)
intraabdominal abscess (Surgical and medical procedures) | 1 (1) | 2 (2) | 0 (0)
hernia (Surgical and medical procedures) | 0 (0) | 4 (4) | 1 (1)
transfusion (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
transient renal insufficiency (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
NSTEMI/STEMI/arrhythmia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
intravenous hydration for hypovolemia (Vascular disorders) | 2 (2) | 9 (9) | 1 (1)
pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No